CLINICAL TRIAL: NCT05742373
Title: Investigating the Role of Fasted Exercise on Improving Cardiometabolic Health; a Potential Mediatory Role of Sirtuins
Brief Title: Role of Fasted Exercise on Improving Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Collaborators: European Society for Clinical Nutrition and Metabolism (Other)
Responsible Party: Principal Investigator, Adora Yau, Senior Lecturer, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FastExTrainESPEN2022
Record Dates: First submitted 2023-01-27; First posted 2023-02-24 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity
Keywords: Cardiovascular disease; Diabetes Mellitus; Obesity; Cardiometabolic health; Exercise; Fasted; Sirtuins
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasted exercise (Experimental): Exercise training in the fasted state
  Interventions: Other: Exercise training in the fasted state
- Fed exercise (Active Comparator): Exercise training in the fed state
  Interventions: Other: Exercise training in the fed state
- Control (No Intervention): No exercise training

INTERVENTIONS:
Other: Exercise training in the fasted state — Four weeks of moderate intensity cycling exercise, three times a week without eating breakfast meal
  Arms: Fasted exercise
Other: Exercise training in the fed state — Four weeks of moderate intensity cycling exercise, three times a week, after eating breakfast meal
  Arms: Fed exercise

SUMMARY:
The aim of this randomised control trial is to investigate the role of fasted exercise on cardiometabolic health. Participants will be assigned to one of three conditions, fasted exercise, fed exercise and control (no exercise). Participants in the exercise groups will complete four weeks of moderate intensity cycling exercise, three times per week, either in the fasted or fed state according to their group assignment. Experimental trials involving anthropometric and cardiometabolic disease risk factor measurements as well as metabolic responses to a subsequent meal ingestion following exercise will be compared pre-intervention and post intervention.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of fasted exercise on cardiometabolic health and the potential mediatory role of sirtuins.

The objectives are to investigate:

1. The effect of a single bout of fasted exercise on acute metabolic responses following a high fat meal.
2. The effect of four weeks of fasted exercise training on cardiovascular and metabolic disease risk factors.
3. The effect of four weeks of fasted exercise training on circulating levels and subcutaneous adipose tissue gene expression of SIRT1, SIRT3 and SIRT6.

A randomised control trial will be conducted with volunteers allocated under the conditions of a) no exercise (control), b) fasted exercise training (FASTEX) and c) fed exercise training (FEDEX). The pre- and post-intervention visits will consist of 50 minutes of cycling at a moderate exercise intensity for both the FASTEX and FEDEX groups. The control group would not perform any exercise. The FASTEX group will perform the exercise in the fasted state, whilst the FEDEX and control groups will be fed a standardised breakfast meal one hour in advance of the exercise period. Following the exercise period, the participants will be fed a high fat meal and metabolic responses to the meal will be measured for four hours. Multiple blood samples will be obtained as well as a sample of subcutaneous adipose (fat) tissue. The FASTEX and FEDEX groups will then complete four weeks of moderate intensity continuous exercise training, either fasted or fed according to their group, on three days per week whilst the control group will maintain their normal sedentary lifestyle. All participants will return to the laboratory for post-intervention testing at the end of the four weeks with the same protocols and measurements as the pre-intervention testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Non-smokers
* Physically inactive (partake in no more than one exercise session per week on average)
* Body mass index >18.5 kg/m2
* Healthy as assessed by medical screening questionnaire
* Prior recipient of local anaesthetic with no known adverse effects, no known hypersensitivity or no other health issue that may constrain the administration of lidocaine hydrochloride
* Free from musculoskeletal injury and able to perform cycling exercise
* Capacity to give informed consent

Exclusion Criteria:

* Regular exerciser
* BMI < 18.5 kg/m2
* Pregnant
* Allergy or intolerances to test meal products/ingredients (such as wheat or dairy products).
* Recent major body weight change (+/- 3 kg in the past month)
* Known hypersensitivity to Lidocaine Hydrochloride
* Cardiovascular disease - complete heart block or hypovolaemia
* Adam's-Stokes Syndrome
* Wolff-Parkinson-White Syndrome
* Porphyria
* Epilepsy
* Myasthenia Gravis
* Other chronic medical condition or diagnosis including respiratory (eg asthma), endocrine, cardiovascular, neuromuscular disorders.
* Taking medications or receiving treatment that may constrain the administration of lidocaine or local anaesthesia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Changes in circulating concentrations of key metabolic markers following a high fat lunch meal | 9 blood samples collected at pre-meal ingestion then every 30 min after ingestion for four hours
  Serum concentrations of clinical chemistry blood analytes (glucose, triglycerides, cholesterol)
Changes in circulating concentrations of key metabolic markers during the experimental trial day | 12 blood samples collected at 0 (baseline), 75 (pre-exercise), 125 (immediately post-exercise), 155 min (pre-meal ingestion) then every 30 min after ingestion for four hours
  Serum concentrations of clinical chemistry blood analytes (glucose, triglycerides, cholesterol)
Area under the circulating concentration versus time curve (AUC) of key metabolic markers following a high fat lunch meal | 4.5 hours
  Total responses of clinical chemistry blood analytes (glucose, triglycerides, cholesterol)
Changes in cardiovascular and metabolic disease biochemistry risk factors | 4 weeks (pre and post intervention)
  Fasted serum concentrations of clinical chemistry blood analytes (glucose, blood lipids, inflammatory markers)
Changes in cardiovascular disease physiological risk factors | 4 weeks (pre and post intervention)
  Systolic and diastolic blood pressure and calculation of mean arterial pressure using systolic and diastolic values
Changes in concentration of sirtuin molecules | 4 weeks (pre and post intervention)
  Serum concentrations of sirtuins
Changes in sirtuin molecule gene expression | 4 weeks (pre and post intervention)
  Adipose tissue gene expression of sirtuins
Changes in sirtuin molecule tissue expression | 4 weeks (pre and post intervention)
  Adipose tissue expression and cellular localisation of sirtuins

SECONDARY OUTCOMES:
Changes in cardiovascular and metabolic disease anthropometric risk factors | 4 weeks (pre and post intervention)
  Waist circumference, hip circumference and waist:hip ratio
Change in body composition | 4 weeks (pre and post intervention)
  Body fat percentage measured using bioelectrical impedance analysis
Change in body mass | 4 weeks (pre and post intervention)
  Body mass in kilograms
Change in substrate oxidation during the experimental trial day | 17 measurements at 0 (baseline), 15 (post-breakfast meal period), 45 (30 min post-breakfast meal period), 75 (pre-exercise), every 10 min during exercise, 155 (pre-meal ingestion), then every 30 min for four hours.
  Carbohydrate and fat oxidation through indirect calorimetry
Heart rate response to exercise | At rest before exercise then every 5 min during 50 min cycle exercise
  Heart rate during exercise in the experimental trial using telemetry
Perceived exertion | Every 5 min during 50 min cycle exercise
  Rating of perceived exertion of exercise in the experimental trial using Borg scale
Change in physical activity levels | Daily for 4 weeks
  Physical activity energy expenditure during the intervention period
Change in physical activity duration | Daily for 4 weeks
  Amount of time spent performing physical activity at different intensities (low, moderate, high) during the intervention period
Change in energy intake | Daily for 4 weeks
  Energy intake using weighed food diary record during the intervention period
Change in dietary nutritional intake | Daily for 4 weeks
  Macronutrient (carbohydrate, fat, protein) composition of food intake using weighed food diary record during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Adora Yau, PhD, Principal Investigator — Manchester Metropolitan University; Gethin Evans, PhD, Study Director — Manchester Metropolitan University
Locations (1):
- Manchester Metropolitan University, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Planned communication of group results at a scientific conference. Planned publication in a scientific peer reviewed journal. Participant level data is not expected to be available as this complies with the conditions of the ethical approval granted for this study.